CLINICAL TRIAL: NCT04275336
Title: Pharmacological and Non-pharmachological Interventions in Management of Peripheral Venipuncture Related Pain: a Randomized Clinical Trial
Brief Title: Pharmacological and Non-pharmacological Interventions in Management of Venipuncture Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FNF201829
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Child, Hospitalized
Keywords: Children; venipuncture related pain and stress; EMLA; distraction techniques
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EMLA group (Experimental): The specialist nurse who is to perform IV cannulation determine the puncture site. A thick layer of cream (lidocaine and propiocaine 2.5%/2.5%) will be applied on a 1x1 cm2 area of skin on the cannulation site. The transparent dressing will be left in place for 30 minutes, then remove and clean with a sterile cotton swab. Then nurse performed IV cannulation for them.
  Interventions: Drug: EMLA application
- Distraction group (Experimental): The multiple distractions including toy whistles, cartoon books, a TV showing cartoons, and various electronic products with video games will be provided for the children to choose and play with. They are also taught breathing exercises (i.e. inhaling through the nose for 3 seconds and exhaling for 5 seconds, while they are counting) if they are willing. A play therapist play with the children for 5 min. prior to and throughout the venipuncture procedure.
  Interventions: Behavioral: Distraction techniques
- Combined group (Experimental): both EMLA cream and distraction techniques will be used. EMLA cream will be applied on the pre-puncture site for 30 minutes as the EMLA group, then 5 minutes before the venipuncture, the play therapist encourage them to choose their favorite toys to play with or to learn breathing exercises. During IV cannulation the play therapist will also continue distracting the child with toys.
  Interventions: Other: EMLA cream and distraction techniques

INTERVENTIONS:
Drug: EMLA application — A thick layer of cream (lidocaine and propiocaine 2.5%/2.5%) will be applied on a 1x1 cm2 area of skin on the cannulation site. The transparent dressing will be left in place for 30 minutes, then remove and clean with a sterile cotton swab. Then nurse perform IV cannulation for them.
  Other Names: EMLA cream
  Arms: EMLA group
Behavioral: Distraction techniques — Multiple distractions including toy whistles, cartoon books, a TV showing cartoons, and various electronic products with video games will be provided for the children to choose and play with. They will also be taught breathing exercises (i.e. inhaling through the nose for 3 seconds and exhaling for 5 seconds, while they are counting) if they are willing. A play therapist play with the children for 5 min. prior to and throughout the venipuncture procedure.
  Other Names: Distractions
  Arms: Distraction group
Other: EMLA cream and distraction techniques — both EMLA cream and distraction techniques will be used. EMLA cream will be applied on the pre-puncture site for 30 minutes as the EMLA group, then 5 minutes before the venipuncture, the play therapist encourage them to choose their favorite toys to play with or to learn breathing exercises. During IV cannulation the play therapist will also continue distracting the child with toys.
  Other Names: EMLA cream and distractions
  Arms: Combined group

SUMMARY:
To evaluate whether an integration of pharmacological and non- pharmacological interventions is more effective than either one of intervention in pain reduction during pediatric peripheral venipuncture.

DETAILED DESCRIPTION:
Intravenous infusion is a routing practice of drug administration for hospitalized children.However numerous studies have shown that venipuncture is a major source of pain of children during their hospitalization which can lead to moderate to severe pain and cause fear, stress and anxiety in children if there is no effective pain management.

The current pain relieving methods include pharmacological (i.e. topical anesthetic) and non-pharmnacological (i.e. distraction techniques) interventions. pharmacological There are scarce evidences supporting that a combination of pharmacological and non-pharmacological interventions can enhance children's abilities in coping with their pain and stress during the venipuncture. EMLA cream is a main pharmacological intervention in managing needle-related pain which can penetrate the cuticle and epidermal layer of intact skin, enter the dermis where nerve endings are located, and relieve pain. However pharmacological interventions have proven inadequate in mitigating pain and stress.The main non-pharmacological alternatives is distraction techniques. There are extremely limited data studies on merging pharmacological and non-pharmacological interventions to compensate for each other's inadequacies. Hence, this study aimed to evaluate the effect of combining both topical anesthetic and distraction techniques in comparison with either of the interventions applied singly.

This study adopts a randomized, blind, controlled intervention trial. Participants will be randomly assigned to three groups: EMLA group, Distraction group and Combined group (EMLA cream plus distraction techniques). The outcomes will be measured by self-reported pain, parent-reported pain and observer-reported pain. Salivary cortisol level will be measured by the ultra sensitive Cortisol Saliva ELISA Assay Kit. Other physiological metrics like heart rate, SpO2, and other intravenous cannulation factors will be rated and recorded.

ELIGIBILITY:
Inclusion Criteria:

Children aged 3-16 years who receive first peripheral intravenous puncture during hospitalization.

Exclusion Criteria:

1. Emergency peripheral intravenous puncture.
2. Allergic history for lidocaine cream.
3. Presence of cognitive impairment, hearing impairment or visual impairment.
4. Children who were discharged from the hospital after participating in the experiment but were readmitted due to illness.
5. Refuse to participate in the study.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 354 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu Z, Zhou Y, Xu X, Lin L, Le Q, Gu Y. Pharmacological and non-pharmacological interventions in management of peripheral venipuncture-related pain: a randomized clinical trial. BMC Pediatr. 2023 Feb 3;23(1):58. doi: 10.1186/s12887-023-03855-z. PMID 36737707

RESULTS

PARTICIPANT FLOW:
Groups:
- EMLA Group: Use EMLA cream in the management of peripheral venipuncture pain.
  EMLA cream will be applied on the skin surface of the injection site, 30 minutes prior to procedure. The dosage is 1g per square centimeter.
- Distraction Group: Use distraction techniques (books, toy whistle, cartoon animation, breathing exercises, electronic products）in the management of peripheral venipuncture pain.
  Distraction techniques: A trained play therapist will entertain and distract the child with psychological interventions (books, toy whistle, cartoon animation, breathing exercises, electronic products）starting 5 minutes before the procedure and ending when the child left the room after the procedure. Children can choose one or more.
- Combined Group: Use EMLA cream combined with psychological interventions in the management of peripheral venipuncture pain.
  EMLA combined with distraction techniques: EMLA cream will be applied on the venipuncture site for 30 minutes than play therapist will distract children with the toys(distraction techniques) children choose before 5 minutes and throughout the venipuncture procedure.
Period: Overall Study
Arm/Group | EMLA Group | Distraction Group | Combined Group
Started | 120 | 118 | 116
Completed | 103 | 96 | 100
Not Completed | 17 | 22 | 16
Not completed — First venipuncture failed | 4 | 6 | 5
Not completed — Unscheduled venipuncture | 9 | 13 | 7
Not completed — Failed specimen of saliva | 4 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Distraction Group: Use distraction techniques (books, toy whistle, cartoon animation, breathing exercises, electronic products）in the management of peripheral venipuncture pain.
  Distraction techniques: A trained play therapist will entertain and distract the child with distraction techniques (books, toy whistle, cartoon animation, breathing exercises, electronic products）starting 5 minutes before the procedure and ending when the child left the room after the procedure. Children can choose one or more distraction toys.
- Combined Group: Use EMLA cream combined with distraction toys in the management of peripheral venipuncture pain.
  EMLA combined with distraction techniques: EMLA cream will be applied on the venipuncture site for 30 minutes than play therapist will distract children with the toys(distraction techniques) ,children choose before 5 minutes and throughout the venipuncture procedure.
- Total: Total of all reporting groups
Arm/Group | EMLA Group | Distraction Group | Combined Group | Total
Number analyzed (Participants) | 103 | 96 | 100 | 299
Age, Continuous [Mean (Standard Deviation); unit: Months] | 105.8 (42.1) | 108.4 (40.4) | 104.6 (46.4) | 106.1 (43.0)
Age, Customized [Count of Participants; unit: Participants] — children who were in their 36 to 83 months old are defined as preschool children; children who were in their 84 to 155 months old are defined as school-aged children; children who were in their 156 to 203 months old are defined as adolescents. researchers will collected the baseline characteristics using the demographic questionnaire before any intervention implementation.
  Participants
    Preschool age | 40 | 29 | 42 | 111
    School age | 47 | 49 | 40 | 136
    Adolescence | 16 | 18 | 18 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 45 | 132
  Male | 56 | 56 | 55 | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 100 | 94 | 98 | 292
  Uyghur | 2 | 1 | 1 | 4
  Zhuang | 0 | 1 | 1 | 2
  Miao | 1 | 0 | 0 | 1
  others | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 103 | 96 | 100 | 299
Age [Geometric Mean (Full Range); unit: Months] | 105.8 [36 to 203] | 108.4 [37 to 203] | 104.6 [36 to 203] | 106.1 [36 to 203]

OUTCOME MEASURES:

1. Primary Outcome: Child Self-reported Pain: Wong-Baker Faces Pain Rating Scale
Description: Pain outcomes are assessed by child himself or herself using Wong-Baker Faces Pain Rating Scale. The scale includes 6 facial expressions with correlating numbers of 0(no hurt), 2(hurts little bit), 4(hurts little more), 6(hurts even more), 8(hurts whole lot), 10(hurts worst). Children pick a facial expression, that corresponds with their pain and see a number that matches it. The minimum value is 0 and the maximum value is 10, the higher score means a worse outcome (children having higher level of pain).
Time Frame: Immediately after completing peripheral venipuncture.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- EMLA Group: Use EMLA cream in the management of peripheral venipuncture pain.
  A eutectic mixture of local anesthetics (EMLA) cream containing 25mg lidocaine and 25mg propiocaine per gram will be applied on the skin surface of the injection site, 30 minutes prior to procedure. The dosage is 1g per square centimeter.
- Distraction Group: Use distraction techniques (books, toy whistle, cartoon animation, breathing exercises, electronic products）in the management of peripheral venipuncture pain.
  distraction techniques: A trained play therapist will distract the child with distraction techniques (books, toy whistle, cartoon animation, breathing exercises, electronic products）starting 5 minutes before the procedure and throughout the whole venipuncture procedure. Children can choose one or more distractions techniques.
- Combined Group: Use EMLA cream combined with distraction techniques in the management of peripheral venipuncture pain.
  EMLA with distraction techniques: EMLA cream will be applied on the venipuncture site for 30 minutes than the play therapist will distract children using distraction techniques 5 minutes before and throughout the venipuncture. procedure.
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
score on a scale | 2 [0 to 2] | 2 [0 to 2] | 2 [0 to 2]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.511, Kruskal-Wallis — <0.05; H value = 1.344

2. Primary Outcome: Parents Reported Pain (Outcomes Assessor ): Revised Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale (r-FLACC)
Description: The effectiveness is analyzed by outcomes assessors using r-FLACC via video taken during the procedure. The outcomes assessor is blind for the study design. The r-FLACC is a tool which evaluates pain-related behavior on facial expression, leg movement, activity, cry and consolability. Total score of the scale is summed in range 0 to 10. 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain.the higher scores mean a worse outcome.
Time Frame: Immediately after completing all participants' interventions.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
score on a scale | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.072, Kruskal-Wallis — <0.05; H value = 5.272

3. Primary Outcome: Observer Reported Pain (Parents): Revised Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale (r-FLACC)
Description: Pain outcomes are assessed by parents using the r-FLACC scale. The r-FLACC is a tool which evaluates pain-related behavior on facial expression, leg movement, activity, cry and consolability. Total score of the scale is summed in range 0 to 10. 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain. The higher scores means a worse outcome
Time Frame: Immediately after completing peripheral venipuncture.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
score on a scale | 1 [0 to 2] | 1 [0.25 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.906, Kruskal-Wallis — <0.05; H value = 0.198

4. Secondary Outcome: Concentration of Salivary Cortisol
Description: Physiological stress levels are measured by means of salivary cortisol as an indicator. The salivary samples (1-2 milliliter) are taken with sterile collection devices immediately after children reporting pain score. The salivary samples are immediately stored at -20℃ freezer. Cortisol levels are determined by human salivary cortisol ELISA Kit (Jianglai, Shanghai, China). This si no cut-off score and the higher scores means a worse outcomes
Time Frame: Immediately after children reporting pain score
Measure: Median (Inter-Quartile Range); unit: percentage of salivary cortisol
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
percentage of salivary cortisol | 35.47 [27.05 to 43.225] | 32.02 [24.525 to 40.7875] | 37.7 [28.01 to 44.645]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.035, Kruskal-Wallis — <0.05; H value = 6.679

5. Secondary Outcome: Heart Rate
Description: Evaluate the physiological response (heart rate) caused by peripheral intravenous puncture. A portable recording pulse oximeter is connected to children's index finger. Heart rate (beats per minute) is measured and recorded.
Time Frame: During the peripheral intravenous insertion procedure.
Measure: Mean (Standard Deviation); unit: beat per minute
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
beat per minute | 104.02 (19.5) | 102.49 (17.72) | 103.65 (20.17)
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.844, ANOVA — <0.05; Mean Difference (Final Values) = 0.170

6. Secondary Outcome: Pulse Oximetry Saturation
Description: Evaluate the physiological response (pulse oximetry saturation) secondary to peripheral intravenous puncture. A portable recording pulse oximeter is connected to children's index finger. Pulse oximetry saturation（percentage）is measured and recorded.
Time Frame: During the peripheral intravenous insertion procedure.
Measure: Median (Inter-Quartile Range); unit: percent of oxyhemoglobin
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
percent of oxyhemoglobin | 98 [97 to 100] | 98 [97 to 100] | 99 [97 to 100]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.438, Kruskal-Wallis — <0.05; H value = 1.651

7. Secondary Outcome: Retaining Time of Intravenous Cannula
Description: Time (hours) from needle insertion to remove.
Time Frame: When the needle is removed.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
hours | 15 [5 to 47] | 15 [5 to 44] | 21 [5 to 52]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.843, Kruskal-Wallis — <0.05; H value = 0.341

8. Secondary Outcome: Venipuncture Duration
Description: record how long is children's first venipuncture duration
Time Frame: During children's first venipuncture
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | EMLA Group | Distraction Group | Combined Group
Number analyzed (Participants) | 103 | 96 | 100
seconds | 83 [70 to 100] | 83 [70 to 96] | 85.5 [74 to 98.75]
Statistical Analysis 1: Comparison: EMLA Group vs Distraction Group vs Combined Group; Test type: Other; p = 0.440, Kruskal-Wallis — <0.05; Median Difference (Final Values) = 1.642

ADVERSE EVENTS:
Time Frame: Throughout the venipuncture procedure and follow-up during children's whole hospitalization, up to 24h
Groups:
- Combined Group: Use EMLA cream combined with distraction in the management of peripheral venipuncture pain.
  EMLA combined with distraction techniques: EMLA cream will be applied on the venipuncture site for 30 minutes than play therapist will distract children with the toys(distraction techniques) children choose before 5 minutes and throughout the venipuncture procedure.
Arm/Group | EMLA Group | Distraction Group | Combined Group
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/96 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/96 | 0/100
Other Adverse Events (participants affected / at risk) | 0/103 | 0/96 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04275336/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT04275336/ICF_001.pdf